CLINICAL TRIAL: NCT04857268
Title: Diagnostic Validation of Wearable Continuous ECG Monitoring Patch, ATP-C120, in High Risk Patients for New-onset Atrial Fibrillation
Brief Title: Diagnostic Validation of Wearable ECG Monitoring Patch, ATP-C120
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Seoul National University Bundang Hospital (Other)
Collaborators: Kyungpook National University Hospital (Other)
Responsible Party: Principal Investigator, Chang-Hwan Yoon, Professor, Seoul National University Bundang Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: B-2009/634-003
Record Dates: First submitted 2021-04-20; First posted 2021-04-23 (Actual); Last update posted 2021-04-26 (Actual); Status verified 2021-04

CONDITIONS: Atrial Fibrillation New Onset
Keywords: Arrhythmia; Atrial Fibrillation; Wearable Electronic Device
MeSH Terms: conditions — Arrhythmias, Cardiac; Atrial Fibrillation

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- ATP-C120 application (Experimental): ATP-C120 will be applied to the high patients for new-onset atrial fibrillation
  Interventions: Device: wearable continuous ECG monitoring patch, ATP-C120

INTERVENTIONS:
Device: wearable continuous ECG monitoring patch, ATP-C120 — ATP-C120 is a novel, single-lead ECG monitoring device which can continuously monitor the ECG signal as long as 14 days (11 days if the device is connected to the smartphone via Bluetooth) when attached to skin adjacent to the heart of patients. It weighs about 8.3 g, with a size of 84 × 39 × 8.3 mm.
  When the device is attached to the patient, several predefined methods were utilized to prevent the occurrence of noise or signal loss. First, the skin was cleansed and disinfected using a 70% ethanol solution. Skin hair was removed if needed. Then the protection film was removed from the patient-side surface of the device. The device is placed at the left 3rd intercostal space 45 degrees tilted toward the inside.

SUMMARY:
A new wearable patch-type device, ATP-C120 (ATsens, Seongnam, Korea) is a novel, single-lead ECG monitoring device and can continuously monitor the ECG signal for upto 11 days. This study is designed to experiment its diagnostic capability of new-onset atrial fibrillation in high risk patients. Several studies reported that validated CHA2DS2-VASc score has high performance in predicting new-onset atrial fibrillation and there are over 10 percent of new-onset atrial fibrillation in patients whose calculated CHA2DS2-VASc scores are ≥ 2. Thus, through this study, the investigators sought to evaluate the validation of early detection of new-onset atrial fibrillation by ATP-C120.

DETAILED DESCRIPTION:
The prevention of stroke associated with atrial fibrillation is a leading global health concern. This devastating event is largely preventable with anticoagulant therapy. Therefore, the early detection and accurate diagnosis of arrhythmia are crucial for prevention of adverse outcome. However, because atrial fibrillation is often intermittent and mostly asymptomatic, it is difficult to capture an excise event.

Conventional electrocardiogram (ECG) monitoring devices including multi-lead portable ECG monitoring device, event-detection monitoring device, and implantable ECG monitoring device are useful for early detection of atrial fibrillation, but these devices have various drawbacks such as requirement of multiple out-patient visits and need of invasive implantation of devices.

A new wearable patch-type device, ATP-C120 (ATsens, Seongnam, Korea) is a novel, single-lead ECG monitoring device and can continuously monitor the ECG signal for upto 11 days. It has recently demonstrated its diagnostic capability and safety compared to the conventional ECG monitoring systems . Yet, it has not widely used in real-world. So, this study is designed to experiment its diagnostic capability of new-onset atrial fibrillation in high risk patients. Several studies reported that validated CHA2DS2-VASc score has high performance in predicting new-onset atrial fibrillation and there are over 10 percent of new-onset atrial fibrillation in patients whose calculated CHA2DS2-VASc scores are ≥ 2. Thus, through this study, the investigators sought to evaluate the validation of early detection of new-onset atrial fibrillation by ATP-C120.

ELIGIBILITY:
Inclusion Criteria:

1. patients who provide written and informed consent to participate
2. patients whose calculated CHA2DS2-VASc score is ≥ 2

Exclusion Criteria:

1. subjects previously diagnosed with atrial fibrillation
2. subjects implanted pacemaker, cardioverter-defibrillator, or any electrical devices
3. subjects had skin problems such as allergic contact dermatitis
4. female patients who are pregnant, or lactating status.

Min Age: 19 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 320 (Estimated)
Dates: Start 2020-11-13 (Actual); Primary Completion 2022-12-31 (Estimated); Study Completion 2023-12-31 (Estimated)

PRIMARY OUTCOMES:
Rate of new-onset atrial fibrillation | 11 days
  new-onset atrial fibrillation recognized by ATP-C120 patch device

SECONDARY OUTCOMES:
Rate of new-onset atrial fibrillation | 6 month
  new-onset atrial fibrillation recognized by conventional ECG monitoring device

CONTACTS AND LOCATIONS:
Overall Officials: Chang-Hwan Yoon, MD.,Ph.D., Principal Investigator — Seoul National University Bundang Hospital
Locations (2):
- South Korea (2):
  - Seoul National Universtiy Bundang Hospital, Seongnam-si, Gyeonggi-do
  - Kyungpook National University Hospital, Daegu

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Choi W, Kim SH, Lee W, Kang SH, Yoon CH, Youn TJ, Chae IH. Comparison of Continuous ECG Monitoring by Wearable Patch Device and Conventional Telemonitoring Device. J Korean Med Sci. 2020 Nov 16;35(44):e363. doi: 10.3346/jkms.2020.35.e363. PMID 33200590
- [Result] Gladstone DJ, Spring M, Dorian P, Panzov V, Thorpe KE, Hall J, Vaid H, O'Donnell M, Laupacis A, Cote R, Sharma M, Blakely JA, Shuaib A, Hachinski V, Coutts SB, Sahlas DJ, Teal P, Yip S, Spence JD, Buck B, Verreault S, Casaubon LK, Penn A, Selchen D, Jin A, Howse D, Mehdiratta M, Boyle K, Aviv R, Kapral MK, Mamdani M; EMBRACE Investigators and Coordinators. Atrial fibrillation in patients with cryptogenic stroke. N Engl J Med. 2014 Jun 26;370(26):2467-77. doi: 10.1056/NEJMoa1311376. PMID 24963566
- [Result] Go AS, Hylek EM, Phillips KA, Chang Y, Henault LE, Selby JV, Singer DE. Prevalence of diagnosed atrial fibrillation in adults: national implications for rhythm management and stroke prevention: the AnTicoagulation and Risk Factors in Atrial Fibrillation (ATRIA) Study. JAMA. 2001 May 9;285(18):2370-5. doi: 10.1001/jama.285.18.2370. PMID 11343485
- [Result] Hart RG, Pearce LA, Aguilar MI. Meta-analysis: antithrombotic therapy to prevent stroke in patients who have nonvalvular atrial fibrillation. Ann Intern Med. 2007 Jun 19;146(12):857-67. doi: 10.7326/0003-4819-146-12-200706190-00007. PMID 17577005
- [Result] Potpara TS, Lane DA, Lip GY. Optimizing stroke prevention in atrial fibrillation: better adherence and compliance from patients and physicians leads to better outcomes. Europace. 2015 Apr;17(4):507-8. doi: 10.1093/europace/euv041. No abstract available. PMID 25833879
- [Result] Waks JW, Buxton AE. Risk Stratification for Sudden Cardiac Death After Myocardial Infarction. Annu Rev Med. 2018 Jan 29;69:147-164. doi: 10.1146/annurev-med-041316-090046. PMID 29414264
- [Result] Healey JS, Connolly SJ, Gold MR, Israel CW, Van Gelder IC, Capucci A, Lau CP, Fain E, Yang S, Bailleul C, Morillo CA, Carlson M, Themeles E, Kaufman ES, Hohnloser SH; ASSERT Investigators. Subclinical atrial fibrillation and the risk of stroke. N Engl J Med. 2012 Jan 12;366(2):120-9. doi: 10.1056/NEJMoa1105575. PMID 22236222
- [Result] Camm AJ, Corbucci G, Padeletti L. Usefulness of continuous electrocardiographic monitoring for atrial fibrillation. Am J Cardiol. 2012 Jul 15;110(2):270-6. doi: 10.1016/j.amjcard.2012.03.021. Epub 2012 Apr 12. PMID 22503584
- [Derived] Kwun JS, Lee JH, Park BE, Park JS, Kim HJ, Kim SH, Jeon KH, Cho HW, Kang SH, Lee W, Youn TJ, Chae IH, Yoon CH. Diagnostic Value of a Wearable Continuous Electrocardiogram Monitoring Device (AT-Patch) for New-Onset Atrial Fibrillation in High-Risk Patients: Prospective Cohort Study. J Med Internet Res. 2023 Sep 18;25:e45760. doi: 10.2196/45760. PMID 37721791